CLINICAL TRIAL: NCT07101523
Title: Using Technologies to Promote HEalthy Lifestyles in Adolescents With Intellectual Disabilities
Acronym: IDHEAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: University of Technology Munich (Unknown)
Responsible Party: Principal Investigator, Borja Sañudo, Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDHEAPP_101134252
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-01

CONDITIONS: Intellectual Disabilities (F70-F79); Down Syndrome (DS); Autism Disorder
Keywords: Intellectual Disabilities; Physical Activity; Sedentary Behavior; mHealth; Health Behavior Change; Health Promotion; Lifestyle Intervention
MeSH Terms: conditions — Intellectual Disability; Down Syndrome; Autistic Disorder; Motor Activity; Sedentary Behavior | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: This study followed a multicenter, randomized controlled trial (RCT) design and was conducted in two European cities: Rome (Italy) and Rijeka (Croatia). Participants were stratified by site and randomly assigned to either an experimental group, which received a gamified mHealth-based intervention aimed at improving physical activity and eating habits, or to a control group, which continued with their usual routines without intervention. In Rome, the sample included only individuals with Down syndrome, while in Rijeka the participants had mild to moderate intellectual disabilities without comorbid Down syndrome. Randomization was carried out using a computer-generated sequence, and the allocation was concealed until the moment of assignment. All procedures complied with the ethical standards of the institutional research committees and adhered to the Helsinki Declaration. Informed consent was obtained from participants or their legal representatives.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the behavioral mHealth intervention, participants and intervention facilitators could not be blinded to group allocation. However, outcome assessors and data analysts were masked to group assignments to minimize potential bias in data collection and analysis. Additionally, caregivers and teachers involved in routine support were not informed of specific hypotheses or group distinctions to reduce influence on participant behavior.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention (Experimental): The intervention was carried out over a period of 8 consecutive weeks and was delivered through a mobile application specifically developed for this project, called IDHEApp, which incorporated gamification elements to enhance user engagement and motivation. Participants in the experimental group received a structured mHealth-based program aimed at promoting healthier behaviors in three primary domains: physical activity, sedentary behavior reduction, and dietary improvement. Objective data on physical activity and sedentary behavior were collected using a smartwatch device (Fitbit Versa 3), which was worn by all participants in both the experimental and control groups throughout the study. However, only participants in the experimental group received a daily personalized behavioral challenge targeting one of the following domains:
  1. Increasing physical activity (e.g., "Walk an additional 1,000 steps today");
  2. Reducing sedentary behavior (e.g., "Stand up and move for at least 5 minu
  Interventions: Behavioral: mHealth
- Control (No Intervention): The control group, in contrast, received no intervention and continued with their usual routines without additional support or monitoring beyond the baseline and post-intervention assessments.

INTERVENTIONS:
Behavioral: mHealth — The intervention was carried out over a period of 8 consecutive weeks and was delivered through a mobile application specifically developed for this project, called IDHEApp, which incorporated gamification elements to enhance user engagement and motivation. Participants in the experimental group received a structured mHealth-based program aimed at promoting healthier behaviors in three primary domains: physical activity, sedentary behavior reduction, and dietary improvement. Objective data on physical activity and sedentary behavior were collected using a smartwatch device (Fitbit Versa 3), which was worn by all participants in both the experimental and control groups throughout the study. However, only participants in the experimental group received a daily personalized behavioral challenge targeting one of the following domains:
  1. Increasing physical activity (e.g., "Walk an additional 1,000 steps today");
  2. Reducing sedentary behavior (e.g., "Stand up and move for at least 5 minut
  Arms: Lifestyle intervention

SUMMARY:
IDHEApp will implement various educational technology tools and work with the families, teachers and caregivers to increase physical activity (PA) and improve healthy eating. Due to the current COVID-19 pandemic restrictions, the use of innovative digital technology can contribute not just to distance learning but also to support families and students in remote. However, both healthy habits and technologies are insufficiently addressed in the population with IDD. These needs are in line with the following objectives of the Erasmus+ programme: a) Inclusion and diversity in all fields of education, training, youth and sport; b) Addressing digital transformation through development of digital readiness, resilience and capacity, and c) Encouraging the participation in sport and physical activity.

Educators will find innovative possibilities and the right instruments that will enable them to fulfil their potential through innovative online education & learning & training skills module for lifestyle promotion and others available on the app. Furthermore, mentors and others health professionals (e.g., nursing etc.) will be equipped with knowledge and skills on how to use the app to teach practical skills for PA enhancement in an evidence-based way. Consequently, this project will contribute to [specific objectives - SO]:

- Raise awareness of the importance of healthy and active living among young Europeans with intellectual disabilities.

Different workshops and bigger events (i.e., international conference), together with the involvement of numerous participants from the institutions of this consortium will be ensured. Further, a sensitized community will participate through the social networks and the website itself, in the proposed activities.

- Provide digital resources and tools to the partner entities of the exchange to improve lifestyle of young people with intellectual disabilities.

Best Practices to provide high quality, inclusive digital health education with the best educational technology tools and methodology. A website, a mobile app and different electronic guidelines will be delivered.

- Analyze the current state of use and acceptance of technologies as support in the management of health in adolescent with intellectual disabilities.

DETAILED DESCRIPTION:
Young individuals with intellectual disabilities (ID) often exhibit significant challenges in maintaining healthy lifestyle habits, particularly concerning physical activity and nutrition. Current evidence indicates that individuals with ID participate in significantly lower levels of physical activity compared to their typically developing peers, with a substantial proportion not meeting established physical activity guidelines. A recent literature review highlights that adults with ID often exhibit elevated levels of sedentary behaviour, which is associated with increased prevalence of obesity, multimorbidity, and metabolic syndrome. The review emphasizes that sedentary behaviour may contribute to the poor health commonly observed in this population. In addition to insufficient physical activity, dietary patterns among young people with intellectual disabilities often skew towards processed foods high in sugar and fat, further compounding their overall health risks.

Addressing these unhealthy behaviors is critical, as they significantly impact the overall well-being of young individuals with ID. Various strategies have been developed to manage and improve lifestyle-related health outcomes in this population. Interventions focusing on lifestyle modifications commonly emphasize structured exercise programs and nutritional education, aiming to promote sustainable, positive health behaviors. However, traditional intervention approaches often face significant challenges in effectively engaging young people with ID, limiting their long-term impact.

In recent years, mobile health (mHealth) interventions have emerged as innovative tools that leverage technology to enhance physical activity and nutritional habits among young individuals with ID. These digital solutions have demonstrated efficacy in promoting behaviour change through interactive, user-friendly platforms, offering an especially attractive alternative for populations that often encounter barriers in traditional health intervention contexts. Existing studies indicate that mHealth applications can facilitate behaviour modification by providing tailored feedback, goal-setting functionalities, and motivational elements, such as gamification.

Despite the significant promise of mHealth interventions in promoting healthier behaviors, evidence regarding their efficacy specifically among individuals with ID remains scarce. Most existing studies have focused on the general population, with limited research adapting these technologies to the cognitive, social, and communication needs of individuals with ID. Several barriers may limit the effectiveness and scalability of mHealth solutions in this population, including difficulties with digital literacy, limited accessibility features in current applications, lack of caregiver or support system involvement, and challenges related to sustained engagement over time. Consequently, there is a critical need for rigorously designed studies that not only evaluate the effectiveness of mHealth interventions for young individuals with ID, but also systematically address the unique barriers this population faces in accessing and benefiting from such technological innovations. Additionally, a significant gap persists in research that adequately considers the diverse manifestations of intellectual disability (e.g., such as Down syndrome and other neurodevelopmental conditions), leading to an incomplete understanding of the true potential and limitations of mHealth solutions across the full spectrum of cognitive and functional profiles. To date, there are only a limited number of studies specifically exploring the use of mHealth interventions to promote physical activity among individuals with ID. Various initiatives demonstrate the feasibility of integrating digital tools to promote physical activity among individuals with ID, they also present notable limitations. These include small sample sizes and a focus on specific subgroups, which hinder the generalizability of their findings. Furthermore, many of these studies predominantly involved adult participants, leaving a significant gap in research related to younger populations, where early intervention is crucial for fostering long-term healthy behaviors. In response to these gaps, our study aims to conduct a randomized controlled trial (RCT) to assess the effectiveness of mHealth interventions in improving physical activity and nutrition in young individuals with ID. By addressing the unique barriers this population faces in engaging with digital health solutions, our research seeks to provide a more comprehensive and inclusive understanding of how mHealth interventions can positively impact health outcomes during this critical developmental stage. Through this approach, we aim to identify effective strategies for promoting sustainable behavior change in young individuals with ID.

Methods Study Design This study followed a multicenter, randomized controlled trial (RCT) design and was conducted in two European cities: Rome (Italy) and Rijeka (Croatia). Participants were stratified by site and randomly assigned to either an experimental group, which received a gamified mHealth-based intervention aimed at improving physical activity and eating habits, or to a control group, which continued with their usual routines without intervention. In Rome, the sample included only individuals with Down syndrome, while in Rijeka the participants had mild to moderate intellectual disabilities without comorbid Down syndrome. Randomization was carried out using a computer-generated sequence, and the allocation was concealed until the moment of assignment. All procedures complied with the ethical standards of the institutional research committees and adhered to the Helsinki Declaration. Informed consent was obtained from participants or their legal representatives.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intellectual disability
* Being able to follow basic instructions
* Age between 4-30 years old

Exclusion Criteria:

* presence of severe sensory or motor impairments
* medical conditions that contraindicated moderate physical activity
* unable to access an smartphone during the intervention

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Daily step count | From enrollment to the end of treatment at 8 weeks
  was recorded as a proxy for general physical activity volume. This variable captured the total number of steps taken each day

SECONDARY OUTCOMES:
light activity | From enrollment to the end of treatment at 8 weeks
  Periods of low-intensity movement such as slow walking or light household tasks,
Sitting time | From enrollment to the end of treatment at 8 weeks
  Total duration per day spent seated, used as a direct indicator of sedentary behavior
Total sleep time | From enrollment to the end of treatment at 8 weeks
  Sum of all sleep periods in a given night
Children's Physical Activity Questionnaire (CPAQ) | From enrollment to the end of treatment at 8 weeks
  To assess self-reported physical activity and sedentary behavior, the Children's Physical Activity Questionnaire (CPAQ) was administered to participants with the support of caregivers or facilitators when necessary. The CPAQ is a semi-structured, interviewer-administered instrument designed to evaluate the typical weekly frequency and duration of different activity types over the previous 7 days. Although originally developed for children, the CPAQ has been successfully adapted and validated in populations with intellectual and developmental disabilities due to its straightforward language and structure (McQueen et al., 2024).
Sleep quality | From enrollment to the end of treatment at 8 weeks
  Pittsburgh Sleep Quality Index (PSQI) A widely used instrument that assesses sleep quality over a one-month interval. It consists of 19 items grouped into 7 components: a) Subjective sleep quality, b) Sleep latency (time to fall asleep), c) Sleep duration, d) Habitual sleep efficiency, e) Sleep disturbances, f) Use of sleep medication, g) Daytime dysfunction. Each component is scored from 0 to 3, and the sum yields a global score (0-21), with higher scores indicating poorer sleep quality. A global score >5 is considered indicative of poor sleep.
health-related quality of life (HRQoL) | From enrollment to the end of treatment at 8 weeks
  To assess health-related quality of life (HRQoL) in individuals with intellectual disabilities, the study employed the Quality of Life Inventory - Intellectual Disability (QI-Disability). This is a validated, condition-specific instrument designed to capture the multidimensional nature of quality of life in individuals with cognitive impairments, including those with mild to severe intellectual disability (Downs et al., 2019). The QI-Disability evaluates six core domains of HRQoL: a) Physical Health, b) Negative Emotions, c) Positive Emotions, d) Social Participation, e) Interpersonal Relationships and f) Independence. Each item is rated on a 4-point Likert scale ranging from "never" to "always," with higher scores indicating a more favorable quality of life in the respective domain. The QI-Disability has shown robust psychometric properties, including high internal consistency and construct validity, in populations with intellectual disabilities (Downs et al., 2019). Importantly, it

CONTACTS AND LOCATIONS:
Overall Officials: Borja Sañudo, PhD, Principal Investigator — University pof Seville
Locations (1):
- Facultad Ciencias de la Educación, Seville, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that will be shared include de-identified data related to primary and secondary outcomes, such as measures of physical activity (e.g., step counts, activity duration), sleep duration, and nutrition-related behaviors. Only IPD used in the results publication will be shared. No personally identifiable information will be included. Data will be shared in accordance with applicable ethical approvals and data protection regulations. Due to the vulnerability of the study population, access to the IPD will be limited to qualified researchers upon reasonable request and subject to a data sharing agreement that ensures confidentiality and appropriate data use.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data (IPD) will be made available beginning 6 months after publication of the primary results and will remain available for a period of 5 years following publication.
Access Criteria: Access to the de-identified individual participant data (IPD) will be granted to qualified researchers affiliated with academic or non-profit institutions for the purpose of secondary analyses related to intellectual disabilities, mHealth interventions, or health promotion. Requests must include a detailed research proposal, ethical approval or exemption, and a signed data use agreement. All requests will be reviewed by the study steering committee to ensure appropriate use and compliance with data protection regulations.